CLINICAL TRIAL: NCT03912441
Title: Open-label Non-Comparator Multicohort Trial of Pharmacokinetics, Safety And Immunogenicity of BCD-147 (JSC "BIOCAD", Russia) After Single Administration of Escalating Doses in Healthy Volunteers
Brief Title: First-In-Human Study to Evaluate Safety And Pharmacokinetics of Single Escalating Doses of BCD-147 (Bispecific Anti-HER2/HER2 Antibody) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BCD-147-1
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BCD-147 Monotherapy Dose Level 1 (Experimental)
  Interventions: Biological: BCD-147
- BCD-147 Monotherapy Dose Level 2 (Experimental)
  Interventions: Biological: BCD-147
- BCD-147 Monotherapy Dose Level 3 (Experimental)
  Interventions: Biological: BCD-147
- BCD-147 Monotherapy Dose Level 4 (Experimental)
  Interventions: Biological: BCD-147

INTERVENTIONS:
Biological: BCD-147 — Bispecific anti-HER2 monoclonal antibody

SUMMARY:
This is an open-label, phase 1, "3+3 trial" of pharmacokinetics, safety and immunogenicity of BCD-147 (JSC "BIOCAD", Russia) after single administration of escalating doses in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form and the subject's ability to follow the Protocol requirements;
2. Male gender 18-45 years of age inclusively at the signing of the informed consent;
3. Body mass index (BMI) in the normal range (18.0 - 30.0 kg / sq.m.);
4. Left ventricular ejection fraction is at least 55% measured by echocardiography;
5. Volunteer's ability to follow Protocol's procedures;
6. Verified diagnosis: "Healthy" according to standard clinical, laboratory, and instrumental examination methods;
7. Hemodynamic parameters within the normal range: systolic blood pressure (BP) in the range of 90-130 mm Hg., diastolic blood pressure in the range of 60-90 mm Hg., heart rate - 60-90 beats / min;
8. Consent of volunteers and their sexual partners with childbearing potential to use adequate contraception throughout the entire trial period. This includes the use of the 1st barrier method in combination with one of the following: spermicides, intrauterine device / oral contraceptives;
9. Volunteer's ability not to drink alcohol within 24 hours prior to the administration of the drug and throughout the entire trial period.

Exclusion Criteria:

1. Participation in any other clinical trial within 30 days before the signing of the informed consent for this clinical trial;
2. Any condition that prevents a patient from following the Protocol procedures (dementia, neurological or mental disorders, drug/alcohol abuse, etc.);
3. The inability of venous puncture for the collection of blood samples (e.g., due to skin diseases);
4. Any surgical procedures that have been transferred within less than 28 days before the signing of the informed consent or planned within 28 days after completion of study participation;
5. Presence of any disorders that, according to the researcher, may affect the pharmacokinetics and safety of the investigational drug;
6. HBV/HCV/HIV infection, active syphilis;
7. Acute infection or the acute phase of chronic infection within 28 days prior the first dose of the investigational product; Active HBV/HCV/HIV infection, active syphilis;
8. Values of standard laboratory and instrumental indicators that go beyond the limits of laboratory standards adopted in the central laboratory;
9. Use of medicines that have a pronounced effect on hemodynamics, liver function, etc. (barbiturates, omeprazole, cimetidine, etc.) less than 28 days before the signing of informed consent and / or the need to take any medications throughout the entire study (except for the study drug);
10. Regular use and parenteral administration of any drugs, including non-prescription drugs, vitamins and dietary supplements, less than 14 calendar days before the signing of informed consent;
11. Known severe allergy (anaphylaxis or multidrug intolerance);
12. Hypersensitivity to any of the components of BCD-147;
13. Smoking of more than 10 cigarettes per day;
14. Use of more than 10 units of alcohol per week (1 unit of alcohol is equivalent to ½ liter of beer, 200 ml of wine or 50 ml of spirits) or anamnestic information about alcoholism, drug addiction or drug abuse, or positive tests for alcohol and / or psychotropic / narcotic substances during the screening visit;
15. Donation of 450 ml or more of blood or plasma within 60 calendar days prior to the signing of informed consent;
16. Cardiovascular disorders, including hypertension or hypotension;
17. Edema of the lower limbs within 14 days before the signing of the informed consent;
18. A history of clinically significant systemic diseases;
19. Use of intravenous antibiotics within 7 days before the signing of informed consent.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 days
The percentage of volunteers with treatment-emerged adverse events of any grade per NCI CTCAE 5.0 | 28 days
The percentage of volunteers with treatment-emerged adverse events of grade 3 and higher per NCI CTCAE 5.0 | 28 days
The percentage of volunteers with both binding and neutralizing antibodies | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Roman A Ivanov, Study Director — Vice President R&D, JSC BIOCAD
Locations (1):
- Medical Center "Eco-Safety", Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No